CLINICAL TRIAL: NCT03439163
Title: Large Sample Collection for Observation of PD Patients and Healthy Controls
Brief Title: Large Sample PD Patients and Healthy Controls
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: TAOWU-PD
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Neuro-Degenerative Disease
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — no biospecimen was collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PD patients: the entire group underwent MRI scan
  Interventions: Device: MRI scan

INTERVENTIONS:
Device: MRI scan — All participants underwent the MRI scan

SUMMARY:
Resting-state functional magnetic resonance imaging (RS-fMRI) has frequently been used to investigate local spontaneous brain activity in Parkinson's disease (PD) in a whole-brain, voxel-wise manner. To quantitatively integrate these studies, we conducted a coordinate-based meta-analysis on 15 studies that used amplitude of low frequency fluctuation (ALFF) and 11 studies that used regional homogeneity (ReHo). All these ALFF and ReHo studies have compared PD patients with healthy controls. We also performed a validation RS-fMRI study of ALFF and ReHo in a frequency-dependent manner for a novel dataset consisting of PD and healthy controls.

DETAILED DESCRIPTION:
Seed-based d Mapping (formerly Signed Differential Mapping, SDM) software (version 5.141 for Windows) (www.sdmproject.com) was used for meta-analysis.

For the validation, fMRI data were acquired on a 3 Tesla Magnetic Resonance scanner (Trio system; Siemens Magnetom scanner, Erlangen, Germany) with gradient-echo echo-plannar imaging sequences. Whole brain fMRI scanning was carried out. All participants were instructed to keep their eyes closed, relax, remain motionless, not think of anything in particular, and not fall asleep. Foam pads were used to minimize head motion.

ELIGIBILITY:
Inclusion Criteria:

* The PD diagnoses were based on the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria. Patients were assessed using the UPDRS III and Hoehn and Yahr disability scale.

Exclusion Criteria:

* 1. history of head trauma, 2. substance abuse, 3. psychiatric disorder. For healthy controls, additional exclusion criteria included

  1. any history of neuropsychiatric disorders.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PD patients were enrolled from the inpatients and the outptients. Healthy controlls were enrolled using advertisement (media and internet)
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
decreased spontaneous brain activity in PD patients | 06/2015-01/2016
  We found a decreased spontaneous brain activity in left putamen in PD patients

CONTACTS AND LOCATIONS:
Overall Officials: Tao Wu, Principal Investigator — Xuanwu Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Yes
We've already uploaded all the raw data to a repository of GigaScience, and part of data to the NITRC repository, named as "PD RS-fMRI meta and validation". After the current study publish, we will update the sharing information here.
Supporting Information: Study Protocol, SAP
Time Frame: starting one year at least after publication
Access Criteria: We will follow the two repositories' commands to share the data. The demography information will also be shared. Dr. Tao Wu will review the requests which is only used for scientific research.

REFERENCES:
- [Result] Pan P, Zhan H, Xia M, Zhang Y, Guan D, Xu Y. Aberrant regional homogeneity in Parkinson's disease: A voxel-wise meta-analysis of resting-state functional magnetic resonance imaging studies. Neurosci Biobehav Rev. 2017 Jan;72:223-231. doi: 10.1016/j.neubiorev.2016.11.018. Epub 2016 Dec 1. PMID 27916710
- [Result] Pan P, Zhang Y, Liu Y, Zhang H, Guan D, Xu Y. Abnormalities of regional brain function in Parkinson's disease: a meta-analysis of resting state functional magnetic resonance imaging studies. Sci Rep. 2017 Jan 12;7:40469. doi: 10.1038/srep40469. PMID 28079169
- See also: The web site of DPABI software — http://www.rfmri.org/dpabi
- See also: The web site of SDM software — http://www.sdmproject.com